CLINICAL TRIAL: NCT01292434
Title: Lunch in the Bag: Packing More Fruit, Vegetables, Grain in Preschool Sack Lunches
Brief Title: Lunch is in the Bag: Helping Parents Increase Fruit, Vegetables, and Whole Grains in Preschool Sack Lunches
Acronym: LIITB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Deanna Hoelscher, Professor - School of Public Health, Austin Regional Campus, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LitB-UT-01
Record Dates: First submitted 2011-02-03; First posted 2011-02-09 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Dietary Behavior
Keywords: Diet; Obesity; Child Preschool; Treatment Outcome; Body Mass Index; Intervention Studies; Randomized Controlled Trial; Child Day Care Centers; Schools Nursery; Child Care
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lunch in the Bag Intervention (Experimental): Lunch is in the Bag behavioral intervention: Parents receive a behavioral intervention that includes handouts/newsletters sent to parents from the early care and education (ECE) center, classroom activities and projects, an implementation support calendar, and teacher training.
  Interventions: Behavioral: Lunch is in the Bag behavioral intervention
- Control (No Intervention): Parents received no specific nutrition education intervention at the ECE center, other than usual practice.

INTERVENTIONS:
Behavioral: Lunch is in the Bag behavioral intervention — Multi-component behavior-based activities, includes: parent handouts, teacher training, age-appropriate child classroom activities, parent/child activity stations
  Other Names: Lunch is in the Bag; LiitB
  Arms: Lunch in the Bag Intervention

SUMMARY:
Lunch is in the Bag is an intervention designed to increase fruits, vegetables, and whole grains in sack lunches prepared for preschool children. Lunch is in the Bag includes 5 weeks of parent handouts, classroom activities related to topics in the handouts, parent and child activities to reinforce behavioral constructs, and a one week booster 22 weeks later.

The primary study hypothesis is that Lunch is in the Bag will increase fruit, vegetables, and whole grains in sack lunches. Additional hypotheses are that lunches at child care centers where the program is used will have higher dietary quality than centers without the program and that children at the centers where the program is used will have a smaller increase in body mass index than children at centers with the program.

The study will also look at the child's home environment and the childcare center. Hypotheses for this research question include

1. Children at centers with Lunch is in the Bag will have greater frequency of eating fruits, vegetables, and whole grains at home than those at centers without the program.
2. Compared to parents at centers without the program, parents of children at centers with Lunch is in the Bag will have

   1. Greater knowledge, expected benefits, support, intentions, and belief in their ability for packing fruit, vegetables, and whole grain in their child's sack lunch daily.
   2. Availability of fruit, vegetable, and whole grain in the home pantry.
   3. Number of lunches with temperature in the safe range at time of service.

DETAILED DESCRIPTION:
Lunch is in the Bag is a behaviorally-based, multilevel intervention to increase the availability of fruits, vegetables and whole grains in sack lunches for preschool children. The Lunch is in the Bag program was designed to fit within the limited time available for parents at childcare centers, and includes 5 weeks of parent handouts, classroom activities related to topics in the handouts, parent and child activities to reinforce behavioral constructs, and a one week booster 22 weeks later.

The primary aim of this proposal is to determine if Lunch is in the Bag program improves the nutrient composition of sack lunches parents pack for children. The primary hypothesis for this aim:

- At 6-week and 28-week follow-up periods, compared to children's lunches at the comparison centers, children's lunches in the intervention group will, on average, contain more servings of: a) fruit; b) vegetables; c) whole grains.

The secondary hypotheses for this aim:

1. At 6-week and 28-week follow-up periods, compared to children's lunches at the comparison centers, children's lunches at the intervention centers on average will have higher dietary quality relative to the Dietary Reference Intakes (DRI) for energy, dietary fiber, carbohydrate, saturated fat, trans fat, vitamin A, calcium, iron, and zinc.
2. At 28-week follow-up periods, children at intervention centers will have smaller increase in BMI compared to children in comparison centers.

The secondary aim of this study is to examine effects of the intervention on psychosocial, behavioral, and environmental supports in the child's home environment. Hypotheses for this aim:

At 6-week and 28-week follow-up periods,

1. Compared to children at the comparison centers, children at the intervention centers on average will have greater frequency of eating fruits, vegetables, and whole grain foods at home.
2. Compared to parents of children at the comparison centers, parents of children at the intervention centers on average will have greater

   1. Behavioral capability/knowledge, perceived behavioral control/self-efficacy, expected benefits/attitudes, subjective norms/social support, and intentions for packing fruit, vegetable, and whole grain in the child's lunch sack daily.
   2. Amount of parent-child cooperation in lunch packing decisions and behaviors.
   3. Availability of fruit, vegetable, and whole grain in the home pantry.
   4. Number of lunches with temperature in the safe range at time of service.

Additional aims include the evaluation of factors affecting implementation and adaption of the program.

Childcare centers (n=40) that require parents to send sack lunches from home will be randomized to intervention and control groups. Families (n=800) will be enrolled as parent-child dyads comprised of the primary lunch packer and one 3 to 5 year old child per family. Outcome measures will be assessed at (1) baseline, (2) immediately after the five-week intervention (6 weeks), (3) 3 months later immediately before a "booster" activity (23 weeks), and (4) 5 weeks after the booster (28 weeks). Mediation analyses will be guided by the Theory of Planned Behavior (TPB) and Social Cognitive Theory (SCT), with particular attention to the reciprocal influences of the child's eating behavior and the parent's food packing behavior and perceptions of child food preferences. Qualitative and process data collection will be conducted throughout the intervention. Data from this study will enable us to determine the efficacy and feasibility of a parent-based intervention implemented through childcare centers to increase the availability of fruits, vegetables, and whole grains in diets of preschool children. The ultimate goal for this work is the development of new strategies for the promotion of healthy eating practices in children through childcare centers, which will decrease their risk of cancer and other chronic diseases later in life.

ELIGIBILITY:
Inclusion Criteria:

* One parent (or guardian)-child dyad per family
* The parent or guardian member of the dyad is the person primarily responsible for packing the child's lunch and is able to read English language materials written at the 6th grade level
* The child member of the dyad is age 3 to 5 and participates in daily care during a full day that includes the hours when children eat their lunch

Exclusion Criteria:

* None

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1266 (Actual)
Dates: Start 2008-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in fruit, vegetable, whole grain in the lunch sack from baseline to 6 weeks, 22 weeks, and 28 weeks | Baseline, 6 weeks, 22 weeks, 28 weeks
  Servings of fruit, vegetable, whole grain in the lunch sack

SECONDARY OUTCOMES:
Nutrient evaluation of the lunch sack: change in nutrient contents from baseline to 6 weeks, 22 weeks, and 28 weeks | baseline, 6 weeks 22 weeks, 28 weeks
  Nutrient analysis of the contents of all foods in the child's lunch sack
Increase in body mass index from baseline to 28 weeks | baseline, 28 weeks
  Child's body mass index at 28 weeks compared to baseline obtained by direct measure of child's height and weight.
Change in parental psychosocial variables from baseline to 6 weeks, 22 weeks, and 28 weeks | baseline, 6 weeks, 22 weeks, 28 weeks
  Variables measuring parents' behavioral capability/knowledge, perceived behavioral control/self efficacy, expected benefits/attitudes, subjective norms/social support, and intentions for packing fruit, vegetable, and whole grain in the child's lunch sack daily, measured by a parent questionnaire.
Change in food availability at home from baseline to 6 weeks, 22 weeks, and 28 weeks | baseline, 6 weeks, 22 weeks, 28 weeks
  Amount of fruit, vegetable, and whole grain available in the child's house measured by home inventory tool.
Change in measured temperature of foods in the lunch sack from from baseline to 6 weeks, 22 weeks, and 28 weeks | baseline, 6 weeks, 22 weeks, 28 weeks
  Temperature of foods at time of service at the childcare center, as measured by a temperature gun.
Change in nutrition environment at the center from baseline to 6 weeks, 22 weeks, and 28 weeks | baseline, 6 weeks, 22 weeks, 28 weeks
  Childcare center's environment regarding support for children's intake of recommended amounts of energy, fruits, vegetables, and whole grains.

CONTACTS AND LOCATIONS:
Overall Officials: Deanna M Hoelscher, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Margaret E. Briley, PhD, Principal Investigator — University of Texas at Austin; Cindy R. Roberts-Gray, PhD, Principal Investigator — Third Coast Research & Development, Inc.
Locations (2):
- United States (2):
  - University of Texas School of Public Health Austin Regional Campus, Austin, Texas
  - Department of Nutritional Sciences, College of Human Ecology, University of Texas at Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Briley ME, Ranjit N, Hoelscher DM, Sweitzer SJ, Almansour F, Roberts-Gray C. Unbundling outcomes of a multilevel intervention to increase fruit, vegetables, and whole grains parents pack for their preschool children in sack lunches. Am J Health Educ. 2012 May;43(3):135-142. doi: 10.1080/19325037.2012.10599230. Epub 2012 May 1. PMID 23243631
- [Background] Sweitzer SJ, Ranjit N, Calloway EE, Hoelscher DM, Almansor F, Briley ME, Roberts-Gray CR. Examining How Adding a Booster to a Behavioral Nutrition Intervention Prompts Parents to Pack More Vegetables and Whole Gains in Their Preschool Children's Sack Lunches. Behav Med. 2016;42(1):9-17. doi: 10.1080/08964289.2014.935283. Epub 2014 Oct 10. PMID 24971674
- [Background] Sweitzer SJ, Byrd-Williams CE, Ranjit N, Romo-Palafox MJ, Briley ME, Roberts-Gray CR, Hoelscher DM. Development of a Method to Observe Preschoolers' Packed Lunches in Early Care and Education Centers. J Acad Nutr Diet. 2015 Aug;115(8):1249-59. doi: 10.1016/j.jand.2015.03.012. Epub 2015 May 12. PMID 25975458
- [Result] Sharma SV, Rashid T, Ranjit N, Byrd-Williams C, Chuang RJ, Roberts-Gray C, Briley M, Sweitzer S, Hoelscher DM. Effectiveness of the Lunch is in the Bag program on communication between the parent, child and child-care provider around fruits, vegetables and whole grain foods: A group-randomized controlled trial. Prev Med. 2015 Dec;81:1-8. doi: 10.1016/j.ypmed.2015.07.005. Epub 2015 Jul 17. PMID 26190371
- [Result] Romo-Palafox MJ, Ranjit N, Sweitzer SJ, Roberts-Gray C, Hoelscher DM, Byrd-Williams CE, Briley ME. Dietary Quality of Preschoolers' Sack Lunches as Measured by the Healthy Eating Index. J Acad Nutr Diet. 2015 Nov;115(11):1779-88. doi: 10.1016/j.jand.2015.05.017. Epub 2015 Jul 17. PMID 26190228
- [Result] Roberts-Gray C, Briley ME, Ranjit N, Byrd-Williams CE, Sweitzer SJ, Sharma SV, Palafox MR, Hoelscher DM. Efficacy of the Lunch is in the Bag intervention to increase parents' packing of healthy bag lunches for young children: a cluster-randomized trial in early care and education centers. Int J Behav Nutr Phys Act. 2016 Jan 8;13:3. doi: 10.1186/s12966-015-0326-x. PMID 26746876
- [Derived] Romo-Palafox MJ, Ranjit N, Sweitzer SJ, Roberts-Gray C, Byrd-Williams CE, Briley ME, Hoelscher DM. Adequacy of Parent-Packed Lunches and Preschooler's Consumption Compared to Dietary Reference Intake Recommendations. J Am Coll Nutr. 2017 Mar-Apr;36(3):169-176. doi: 10.1080/07315724.2016.1240634. Epub 2017 Jan 12. PMID 28080325
- [Derived] Roberts-Gray C, Sweitzer SJ, Ranjit N, Potratz C, Rood M, Romo-Palafox MJ, Byrd-Williams CE, Briley ME, Hoelscher DM. Structuring Process Evaluation to Forecast Use and Sustainability of an Intervention: Theory and Data From the Efficacy Trial for Lunch Is in the Bag. Health Educ Behav. 2017 Aug;44(4):559-569. doi: 10.1177/1090198116676470. Epub 2016 Nov 17. PMID 27864471
- See also: Project Website — https://sph.uth.edu/research/centers/dell/project.htm?project=8f5592fc-46aa-475f-a414-3ef239c513fe